CLINICAL TRIAL: NCT06194071
Title: Assessment of the Feasibility of a Systematic Multidimensional Evaluation of the Outcome of Head Injury Patients and Their Families. A Single-center Pilot Cohort With Repeated Longitudinal Follow-up
Brief Title: Assessment of the Feasibility of a Systematic Multidimensional Evaluation of the Outcome of Traumatic Brain Injury Patients and Their Relatives.
Acronym: MUST²
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AR_2023_002
Record Dates: First submitted 2023-11-14; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Traumatic Brain Injury
Keywords: Cohort; Pilot Study; Longitudinal follow-up
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Traumatic Brain Injury: Patients with all types of TBI will be recruited (mild, moderate and severe). They mus accept participation in the prolonged follow-up (up to 18 months after the accident). Relatives will also accept to participate. Patients will undergo routine care regarding TBI in our institution. Only the prolonged follow-up and monitoring is proposed which combines remote questionnaire completion, and on-site visits at 3 time-points (6, 12 and 18 months). No on-site visit is proposed for relatives who will fill out questionnaires. However, they may accompany patients during on-sites visits.
  Interventions: Other: Completion of questionnaires and on-site visits during an 18 months follow-up after TBI

INTERVENTIONS:
Other: Completion of questionnaires and on-site visits during an 18 months follow-up after TBI — We will evaluate the same outcomes and use the same questionnaires at 6, 12 and 18 months post-TBI.
  For patients we will evaluate:
  * Functional Outcome (GOS-Extended)
  * Health-related Quality of Life (QOLIBRI)
  * Neurocognitive tests (MoCA)
  * Independence (Barthel Index)
  * Daily issues (BICOQ)
  * Anxiety and depression symptoms (HADS)
  * Medico-economic evaluation (EQ5D-5L)
  For Relatives we will evaluate:
  * Symptoms of anxiety and depression (HADS)
  * The appreciation of the patient's daily issues from their point of view (dedicated Bicoq for relatives)
  * Burden of care (ZARIT)
  Throughout the follow-up we will nest a qualitative research programs which will focus on several aspects:
  * feasibility of such follow-up (6 months is the primary endpoint) defined as the drop-out rate, complete or incomplete completion of scales and their reasons
  * factors that may lead to drop-out or the contrary that solidifies the follow-up

SUMMARY:
The main objective is to assess the feasibility of collecting and implementing a multidimensional evaluation in a sample of patients with a mild to severe traumatic brain injury (TBI) and their relatives, evaluated at 6 months (primary outcome), and at 12 then 18 months post-injury (secondary outcomes).

DETAILED DESCRIPTION:
The study aims to assess the feasibility of collecting multidimensional outcomes of patients with traumatic brain injury, taking into account the patient-relative dyad. However, this multidimensional assessment may pose enormous problems of feasibility during the follow-up: loss of the patient's pathway, moderate acceptance by patients and relatives, difficulties of remote assessment sometimes carried out several times.... All these factors can affect the methodological quality of the evaluation of patient outcomes, with measurement and reporting biases influencing the results of biomedical trials. In order to improve the quality of clinical research in this field, it is therefore essential to fully appreciate the factors that facilitate or, on the contrary, hinder high-quality longitudinal follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU with Glasgow score during initial car ≤ 14 and CT-confirmed head injury
* Patients admitted to ER with Glasgow score during initial care ≤ 15 or concussion and CT-confirmed head injury or displaying clinicalsigns such as headaches or vomiting.

Exclusion Criteria:

* Patients under 18 years of age
* Single patient, without relative or informal caregiver
* Non-French-speaking patient
* Refusal of consent
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population includes patients with mild to severe traumatic brain injury and their relatives (informal caregivers).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Analysis of the feasibility of multidimensional analysis | 6 months
  The number of scales ( GOS-Extended, QOLIBRI, MoCA, BARTHEL INDEX, BICOQ, HADS, EQ5D-5L, ZARIT) entirely completed
Analysis of the feasibility of multidimensional analysis | 6 months
  the number of missing items per scale
Analysis of the feasibility of multidimensional analysis | 6 months
  the number of patients seen at the on-site visit
Analysis of the feasibility of multidimensional analysis | 6 months
  the number of neur-cognitive tests (MoCA) carried out in full
Analysis of the feasibility of multidimensional analysis | 6 months
  Study the reasons of complete/incomplete items rating
Analysis of the feasibility of multidimensional analysis | 6 months
  Study the reasons for drop out of the follow-up

SECONDARY OUTCOMES:
Analysis of the feasibility of multidimensional analysis | 12 and 18 months
  In-depth analysis of the completion of the follow-up at 12 and 18 months by patients and family caregivers
Analysis of engagement and attrition by the dyad | 12 and 18 months
  The outcomes and questionnaires (GOS-Extended, QOLIBRI, MoCA, BARTHEL INDEX, BICOQ, HADS, EQ5D-5L, ZARIT) will be used throughout the study
Evolution over time of the outcome | 18 months
  Modification in functional outcomes assessed by GOS-Extended during the follow-up
Evolution over time of the outcome | 18 months
  Changes in health-related quality of life outcomes assessed by QOLIBRI during the follow-up
Evolution over time of the outcome | 18 months
  Modification in functional outcomes assessed by Barthel Index during the follow-up
Evolution over time of the outcome | 18 months
  Changes in MoCA neurocognitive test scores during the follow-up
Evolution over time of the outcome | 18 months
  Changes in the results of the BICOQ survey evaluating awareness of issues in day-to-day life during the follow-up
Evolution over time of the outcome | 18 months
  Modification of mood disorder questionnaire results evaluated by HADS during follow-up
Evolution over time of the outcome | 18 months
  Modification of the medico-economic progress assessment using EQ5D-5L questionnaire results during follow-up
Prognostic models | 18 months
  Elaborate original predictive models between the acute phase of in-hospital TBI management. Collection of routine data during in-hospital management

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided